CLINICAL TRIAL: NCT01736631
Title: Cognitive Behavioural Therapy for Social Phobia in People With Bipolar Disorder: A Pilot Study
Brief Title: Cognitive Behavioural Therapy for Social Phobia in People With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBTSPBD-001
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2017-06

CONDITIONS: Social Phobia; Bipolar Disorder
Keywords: social phobia; bipolar disorder; cognitive behavioural therapy
MeSH Terms: conditions — Phobia, Social; Bipolar Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive behavioural therapy (Experimental): Cognitive behavioural therapy for social phobia in people with bipolar disorder
  Interventions: Behavioral: Cognitive behavioural therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy (CBT) — The CBT intervention will follow the model of social phobia by Clark & Wells (Clark & Wells, 1995; Clark, 2005). The main elements of CBT for social phobia include reducing self-focus, dropping safety behaviours, and testing negative cognitions.

SUMMARY:
We are doing this study to find out how well cognitive behavioural therapy for social phobia works in people with bipolar disorder, who also have social phobia.

DETAILED DESCRIPTION:
Social phobia is a very prevalent anxiety disorder in people with bipolar disorder and is associated with adverse outcomes. Yet, social phobia is treatable by cognitive behavioural therapy or antidepressant medication. As antidepressants are often contra-indicated in people with bipolar disorder, cognitive behavioural therapy is the likely first choice treatment for social phobia in this population. However, people with bipolar disorder were excluded from previous clinical trials on treatment of social phobia. Our aim is to evaluate the acceptability and to provide a rough estimate of efficacy of cognitive behavioural therapy protocol for social phobia in people with bipolar disorder in a systematic case series. We will also prepare pilot data for evaluating the impact of treatment of comorbid social phobia on the long-term course of bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of bipolar disorder I or II according to DSM-IV criteria and established in a structured interview
* Bipolar disorder in remission for at least 12 weeks; defined as absence of depressive or manic episode according to DSM-IV criteria established in a structured interview and confirmed by Montgomery-Åsberg Depression Rating Scale score ≤ 12 and Young Mania Rating Scale score ≤ 7
* Stable medication regime for at least 4 weeks prior to commencing CBT
* Current diagnosis of social phobia according to DSM-IV criteria and established in a structured interview, including duration of social phobia of at least 6 months irrespective of age.
* Social phobia is one of the primary complains (when bipolar disorder is in remission), justifying a therapeutic focus on this disorder.
* Ability and willingness to consent to treatment
* Ability to speak and write English

Exclusion Criteria:

* Current substance use disorder
* A previous adequate course of CBT for social phobia (at least 8 sessions) delivered by a trained therapist
* Currently receiving any psychological therapy
* Cognitive impairment that would preclude psychological therapy
* Actively suicidal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Acceptability of cognitive behavioural therapy for comorbid social phobia in bipolar disorder | up to end of treatment (20 weeks)
  Acceptability of cognitive behavioural therapy for comorbid social phobia in bipolar disorder will be assessed as proportion of offered sessions attended
Change on the Social Phobia Inventory (SPIN) | Baseline and end of treatment (20 weeks)

SECONDARY OUTCOMES:
Change on the Liebowitz Social Anxiety Scale Scale Self-Report; Social Phobia Scale & Social Interaction Anxiety Scale; Social Phobia and Anxiety Inventory | Baseline and end of treatment (20 weeks)
Presence/absence of the social phobia diagnosis | Baseline and end of treatment (20 weeks)
  Presence/absence of the social phobia diagnosis as established by Structured Clinical Interview for DSM Disorders
Depression symptom change | Baseline and end of treatment (20 weeks)
  Depression symptom change as established by the Montgomery-Åsberg Depression Rating Scale and Beck Depression Inventory II
Mania symptom change | Baseline and end of treatment (20 weeks)
  Change in symptoms of mania as established by the Young Mania Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pavlova, PhD DClinPsy, Principal Investigator — Capital Health, Canada
Locations (1):
- Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia, Canada